CLINICAL TRIAL: NCT04060147
Title: A Proof-of-Concept, Open-Label Study Evaluating the Safety and Tolerability of Cilofexor in Subjects With Primary Sclerosing Cholangitis (PSC) and Compensated Cirrhosis
Brief Title: Safety and Tolerability of Cilofexor in Participants With Primary Sclerosing Cholangitis (PSC) and Compensated Cirrhosis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study enrollment was terminated early by the sponsor due to recruitment challenges.
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-428-5443
Record Dates: First submitted 2019-08-15; First posted 2019-08-16 (Actual); Results first posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2022-08

CONDITIONS: Primary Sclerosing Cholangitis; Compensated Cirrhosis
MeSH Terms: conditions — Cholangitis, Sclerosing | interventions — cilofexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cilofexor (Experimental): Participants will receive escalating doses of cilofexor 30 mg, 60 mg, and 100 mg.
  Interventions: Drug: Cilofexor

INTERVENTIONS:
Drug: Cilofexor — Tablets administered orally once daily
  Other Names: CILO; GS-9674

SUMMARY:
The primary objective of this study is to assess the safety and tolerability of escalating doses of cilofexor (CILO) in participants with primary sclerosing cholangitis (PSC) and compensated cirrhosis.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis PSC based on cholangiogram (magnetic resonance cholangiopancreatography [MRCP], endoscopic retrograde cholangiopancreatography [ERCP], or percutaneous transhepatic cholangiogram [PTC]) or liver biopsy
* Individuals have evidence of cirrhosis based on historical liver biopsy, abdominal imaging [magnetic resonance imaging (MRI), computed tomography (CT), or Ultrasound], or a screening FibroScan®, enhanced liver fibrosis (ELF)™, or FibroTest®.
* Individual has the following laboratory parameters at the Screening visit, as determined by the central laboratory:

  * Estimated glomerular filtration rate (eGFR) > 60 milliliter/minute (mL/min), as calculated by the Cockcroft-Gault equation
  * Alanine aminotransferase (ALT) ≤ 5 x upper limit of the normal (ULN)
  * Total 2 milligram/deciliter (mg/dL), unless the individual is known to have Gilbert's syndrome or hemolytic anemia
  * International normalized ratio (INR) ≤ 1.4, unless due to therapeutic anticoagulation
  * Platelet count ≥ 75,000/microliter (μL). Individuals with evidence of high-risk esophageal or gastric varices in the opinion of the investigator are excluded
  * Negative anti-mitochondrial antibody

Key Exclusion Criteria:

* Current or prior history of any of the following

  * Decompensated liver disease, including ascites, hepatic encephalopathy (HE), or variceal hemorrhage
  * Liver transplantation
  * Cholangiocarcinoma or hepatocellular carcinoma (HCC).
* Model for End-stage Liver Disease (MELD) score > 12 at Screening, unless due to an alternate etiology such as therapeutic anticoagulation
* Child-Pugh (CP) score > 6 at Screening, unless due to an alternative etiology such as Gilbert's syndrome or therapeutic anticoagulation
* Current moderate to severely active inflammatory bowel disease (IBD) (including ulcerative colitis, Crohn's disease, and indeterminate colitis).

  * Note: Individuals with IBD who currently have an external ostomy bag and/or proctocolectomy are not subject to this exclusion criterion and need not undergo IBD Symptom Severity Assessment.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2021-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (16):
- United States (16):
  - Arizona Liver Health, Chandler, Arizona
  - California Liver Research Institute, Pasadena, California
  - University of California San Francisco, Liver Clinic, San Francisco, California
  - Schiff Center for Liver Diseases/University of Miami, Miami, Florida
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - Indiana University Health University Hospital, Indianapolis, Indiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Minnesota Gastroenterology, PA, Maplewood, Minnesota
  - Northwell Health Center for Liver Diseases and Transplantation, Manhasset, New York
  - University of Rochester Medical Center, Rochester, New York
  - The Liver Institute at Methodist Dallas Medical Center, Dallas, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Bon Secours Richmond Community Hospital, Inc. d/b/a Bon Secours Liver Institute of Richmond, Richmond, Virginia
  - VCU Clinical Research Services Unit (CRSU) [Patient Site Address], Richmond, Virginia
  - University of Washington at Harborview Medical Center, Seattle, Washington
  - Liver Institute Northwest, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Levy C, Caldwell S, Mantry P, Luketic V, Landis CS, Huang J, Mena E, Maheshwari R, Rank K, Xu J, Malkov VA, Billin AN, Liu X, Lu X, Barchuk WT, Watkins TR, Chung C, Myers RP, Kowdley KV. Cilofexor in Patients With Compensated Cirrhosis Due to Primary Sclerosing Cholangitis: An Open-Label Phase 1B Study. Clin Transl Gastroenterol. 2024 Aug 1;15(8):e00744. doi: 10.14309/ctg.0000000000000744. PMID 38976363

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States.
Pre-assignment Details: 18 participants were screened.
Groups:
- Cilofexor: Cilofexor 30 mg tablet orally once daily from Week 1 to Week 4, followed by cilofexor 60 mg (2 X 30 mg) tablets orally once daily from Week 5 to Week 8, followed by cilofexor 100 mg tablet orally once daily from Week 9 to Week 12. Participants received cilofexor for a total duration of 12 weeks.
Period: Overall Study
Arm/Group | Cilofexor
Started | 11
Completed | 10
Not Completed | 1
Not completed — Withdrew consent | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who took at least 1 dose of study drug.
Arm/Group | Cilofexor
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black or African American | 1
  Race: White | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Not Hispanic or Latino | 10
  Ethnicity: Hispanic or Latino | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced Treatment-emergent Adverse Events (TEAEs)
Description: Treatment-emergent adverse events (TEAEs) were either defined any AEs with an onset date on or after the study drug start date and no later than 30 days after permanent discontinuation of study drug or any AEs leading to premature discontinuation of study drug.
Time Frame: First dose date up to 12 weeks plus 30 days
Population: Safety Analysis Set included all participants who took at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cilofexor
Number analyzed (Participants) | 11
percentage of participants | 81.8

2. Primary Outcome: Percentage of Participants Who Experienced Treatment Emergent Serious Adverse Events (SAEs)
Description: A treatment emergent SAE was defined as an event that, at any dose, resulted in the following: death ; life-threatening situation; in-patient hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity; a congenital anomaly/birth defect; a medically important event or reaction: such events may not be immediately life-threatening or result in death or hospitalization but may jeopardize the subject or may require intervention to prevent one of the other outcomes constituting SAEs.
Time Frame: First dose date up to 12 weeks plus 30 days
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cilofexor
Number analyzed (Participants) | 11
percentage of participants | 0

3. Primary Outcome: Percentage of Participants Who Experienced Laboratory Abnormalities
Description: Treatment-emergent laboratory abnormalities are defined as values that increase at least 1 toxicity grade from baseline at any postbaseline time point, up to and including the date of last dose of study drug plus 30 days. Grade 1: mild; Grade 2: moderate; Grade 3: severe; Grade 4: life-threatening.
Time Frame: First dose date up to 12 weeks plus 30 days
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cilofexor
Number analyzed (Participants) | 11
percentage of participants
  Grade 1 | 54.5
  Grade 2 | 36.4
  Grade 3 | 9.1
  Grade 4 | 0

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: Enrollment up to 17 weeks; Adverse Events: First dose date up to 12 weeks plus 30 days
Description: All-cause mortality: All enrolled analysis set included all participants who received a study participant identification number in the study after screening.
  Adverse events: Safety analysis set included all participants who took at least 1 dose of study drug.
Arm/Group | Cilofexor
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 9/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cilofexor (N=11)
Vertigo (Ear and labyrinth disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Defaecation urgency (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 2
Ill-defined disorder (General disorders) | 1
Oedema peripheral (General disorders) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 1
Jaw fracture (Injury, poisoning and procedural complications) | 1
Lip injury (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 2
Menopausal symptoms (Reproductive system and breast disorders) | 1
Oligomenorrhoea (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 8
Rash papular (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2021-01-15): https://cdn.clinicaltrials.gov/large-docs/47/NCT04060147/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-15): https://cdn.clinicaltrials.gov/large-docs/47/NCT04060147/SAP_001.pdf